CLINICAL TRIAL: NCT02630940
Title: Exhaled Breath Condensate Biomarkers and Cough in People With Idiopathic Pulmonary Fibrosis
Brief Title: Exhaled Breath Condensate Biomarkers and Cough in IPF
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: 152379 (113-08-15)
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Idiopathic pulmonary fibrosis sufferers: Male or female idiopathic pulmonary fibrosis (IPF) sufferers over the age of 40, with a confirmed diagnosis of IPF against international guidelines. Patients are devoid of significant other medical, surgical or psychiatric illnesses that may affect respiratory symptoms or disease progression.

SUMMARY:
Analysis of exhaled breath condensate biomarkers and cough severity in patients with idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
This study will aim to investigate the levels of the reactive oxygen species (ROS) 8-isoprostane in idiopathic pulmonary fibrosis patients' exhaled breath condensate (EBC). EBC samples will be collected using RTube, prior to analysis for levels of 8-isoprostane. An acceptability assessment will be performed for this non-invasive method of EBC collection through a non-validated questionnaire.

A regression analysis will then be performed for 8-isoprostane levels against the severity of the patient's cough, assessed through the use of the visual analogue scale for cough (VAS), the King's brief interstitial lung disease questionnaire (KBILD), the Medical Research Council (MRC) dyspnoea scale and the Leicester cough questionnaire. Alongside this an exploratory comparison of cough scores and 8 isoprostane concentration between patients with and without honeycombing and traction bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female above the age of 40
* IPF diagnosed by a multi-disciplinary team meeting following review of clinical history, thoracic high resolution computed tomography (HRCT) and/or surgical lung according to international guidelines

Exclusion Criteria:

* A recognised significant co-existing respiratory disease, defined as a respiratory condition that exhibits a clinically relevant effect on respiratory symptoms and disease progression as determined by the principal investigator following multi-disciplinary discussion. For example, patients with bronchiectasis will only be included if the bronchiectasis is deemed to be traction bronchiectasis as a result of idiopathic pulmonary fibrosis
* Airflow obstruction defined as a forced expiratory volume at one second over forced vital capacity (FEV1/FVC) <60% predicted or a residual volume greater than 120% predicted
* Significant medical ,surgical or psychiatric disease that in the opinion of the patient's attending physician would exhibit a clinically relevant effect on the patient's health related quality of life
* The patient is unable to provide written informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or Female Idiopathic pulmonary fibrosis sufferers over the age of 40, who have been diagnosed in accordance with either a multi-disciplinary review of their clinical history, thoracic high resolution computed tomography and/or surgical lung according to international guidelines
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
8-isoprostane levels | 1 day (Single measurement )
  Used for detection of 8-isoprostane levels in patients' exhaled breath condensate samples

SECONDARY OUTCOMES:
Leicester Cough Questionnaire | 1 day (Single measurement )
  Assessment of patient's cough severity
Kings brief interstitial lung disease questionnaire | 1 day (Single measurement )
  Assessment of patient's cough severity & exercise tolerance
MRC dyspnoea Scale | 1 day (Single measurement )
  Assessment of patient's exercise tolerance
Visual analogue scale for Cough | 1 day (Single measurement )
  Assessment of patient's cough severity
Non-validated acceptability questionnaire | 1 day (Single measurement )
  Assessment of exhaled breath condensate collection method acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Wilson, MD MRCP, Principal Investigator — University of East Anglia; Christopher Atkins, MBBS, Principal Investigator — University of East Anglia; Ashnish Sinha, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom